CLINICAL TRIAL: NCT03974607
Title: Multidisciplinary Training Program for the Promotion of Physical Activity and Other Healthy Habits in Inactive Adolescents
Brief Title: Program to Promote Physical Activity and Healthy Habits in Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Extremadura (Other)
Responsible Party: Principal Investigator, PEDRO ANTONIO SÁNCHEZ MIGUEL, Principal Investigator, University of Extremadura
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: University of Extremadura
Record Dates: First submitted 2019-05-22; First posted 2019-06-05 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-06

CONDITIONS: Activity, Motor
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity (Experimental): Physical Activity Programme (PAP) was planned for the promotion of PA and other healthy habits in inactive adolescents as an agent of change intervention, in which a trained staff actively disseminates effective practices to improve the PA's habits of adolescents.
  Interventions: Behavioral: Physical Activity Program (PAP)
- No Physical Activity (No Intervention): The control group will be selected in a targeted manner according to the availability of the center. You will not be given any information about healthy habits nor will any physical training program be applied to you, so that you do not give indications that may produce a variation of your habitual behavior.

INTERVENTIONS:
Behavioral: Physical Activity Program (PAP) — A Physical Activity Program (PAP) will be carried out. Previously an initial measure will be made to know the little active adolescents. At the end of the PAF a retention measure will be carried out to know the scope and persistence of the variables analyzed. The PAF will be developed with a frequency of three weekly sessions, of 60 minutes, in the period of the intervention, with the exception of weeks in which there is a public holiday, where we will take measures to recover the class. A schedule for the sessions will be set according to the interests of the participants and will be the same for all. During the sessions, basic physical abilities and motor skills will be worked on with playful proposals focused on the improvement of physical and psychosocial parameters. They will always have the same monitor Graduate in Physical Activity and Sports Sciences, which will be responsible for developing the PAF.
  Arms: Physical Activity

SUMMARY:
The main objective of the research project presented is to improve physical activity levels in adolescents who present rates of diagnosed active impairment through the design, development and evaluation of a multidisciplinary intervention program of physical activity to promote healthier lifestyles . This program will follow the principles of the Theory of Self-determination, using Information and Communication Technologies (ICTs), a training plan for monitors, teachers and parents, with the aim of achieving greater adherence to the sports practice of adolescents from Extremadura, with the benefits at a psychosocial, cognitive and biological level that this entails.

DETAILED DESCRIPTION:
The main objective of the research project presented is to improve physical activity levels in adolescents who present rates of diagnosed active impairment through the design, development and evaluation of a multidisciplinary intervention program of physical activity to promote healthier lifestyles . This program will follow the principles of the Theory of Self-determination, using Information and Communication Technologies (ICTs), a training plan for monitors, teachers and parents, with the aim of achieving greater adherence to the sports practice of adolescents from Extremadura, with the benefits at a psychosocial, cognitive and biological level that this entails.

Students of 1st and 2nd year of E.S.O would be part of this project. of different educational centers of the Autonomous Community of Extremadura and the set of professors of the mentioned centers. Through the initial measurement made to 1st and 2nd year students of E.S.O, children who do not perform sufficient physical activity and can be part of the intervention study will be identified. In this way, identified young people who do not perform physical activity or do not reach minimum recommendable values, will be grouped by means of the sampling of random selection by conglomerates in a control group and an experimental group. Overall, the investigatos would expect to have a total of about 240 male and female students, with ages between 11 and 15 years, where about 120 students would be part of the experimental group and another 120 students would form the control group. Indirectly, parents of students and teachers in the area of Physical Education who will collaborate in different activities and events would also participate.

To achieve the objectives of the project, a quasi-experimental methodology would be carried out, with an ABA'-A'' design, formed by a first phase of initial evaluation of the psychosocial and biological variables that the investigators are going to try to optimize, a second phase that would consist of the intervention based on different procedures developed throughout an academic course, a third phase of final evaluation of the different variables that aims to assess the effects of the intervention and the usefulness of the program, and a fourth phase with an extinction measure, aimed at evaluating the stability of the effects caused by the program.

The benefits of this project would be framed in different levels. In the first place, the main benefit would be obtained by the direct recipients of the project, that is, the adolescents who would see their physical activity levels increased with the positive consequences that this entails and with the development of healthier living habits. Secondly, Physical Education teachers could have new methodological and motivational tools to encourage more physical activity among their students; and the parents of these, could value the importance of physical activity and lead an active lifestyle, collaborating from the family environment to promote the objectives of this project.

ELIGIBILITY:
Inclusion Criteria:

* Age: 10 - 16 años
* Nor engaged in regular physical activity > 20 min on > 3 days/week
* Not participating in a weight loss programme
* Provide informed consent by parents, mothers or legal guardians
* Participants must be capable and willing to provide consent, understand exclusion criteria and accept the randomized group assignment.
* Participants must attend at least 80% of the sessions.

Exclusion Criteria:

* Unwillingness to either complete the study requirements or to be randomized into control or training group.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-01-21 (Estimated); Study Completion 2020-07-28 (Estimated)

PRIMARY OUTCOMES:
Perception of physical activity levels | 3 Months
  The levels of PA of adolescents were assessed using a scale designed by the WHO and developed in many countries called the International Physical Activity Questionnaire (IPAQ - A: Hagströmer et al., 2008).
Type of motivation towards sports | 3 Months
  The motivation of the students will be evaluated when doing physical exercise through the versioned Spanish version (BREQ-2: Moreno-Murcia Cervelló, and Martínez, 2007) of the Behavioral Regulation in Exercise Questionnaire (BREQ-3: Wilson Rodgers, Loitz , and Scime, 2006).
Satisfaction of basic psychological needs: scale | 3 Months
  The perception of body image and the desired body image of the students will be analyzed, using the scale of Stunkard, Sørensen, and Schulsinger (1983).
Levels of physical activity | 3 Months
  The level of physical activity will be measured with Actigraph wGT3X-BT accelerometers will be used, with high reliability and information storage capacity.
Body Image Dimensional Assessment | 3 Months
  The dimension of the body image of adolescents will be analyzed with the BIDA questionnaire (Segura-García et al., 2012).
Physical condition | 4 Months
  The physical condition (strength, endurance and agility) will be evaluated by the Alpha Fitness test battery (Ruiz et al., 2011).
Body composition | 4 Months
  The body fat percentage will be assessed through the subscapular and triciple pligues using the Holtain plicter.
Body Mass Index (BMI) | 4 Months
  The BMI of the participants will be evaluated. To do this, all young students will be measured and weighed and the BMI calculated using the following formula: BMI = Weight (Kg) / Height2 (Mt). For this, the Scale (SECA 877), and a Leicester Height Measure brand stadiometer, Marsden Group, will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Antonio Sánchez Miguel, Study Director — University Extremadura; Miguel Angel Tapia Serrano, Principal Investigator — University Extremadura
Locations (1):
- Pedro Antonio Sánchez Miguel, Cáceres, Extremadura, Spain

IPD SHARING:
Plan to Share IPD: No